CLINICAL TRIAL: NCT02503839
Title: Therapeutic Vaccination and Immune Modulation - New Treatment Strategies for the Multidrug-resistant Tuberculosis Pandemic; an Open Label Phase I Clinical Trial of the Therapeutic TB H56:IC31 Vaccine and Cyclooxygenase-inhibitors
Brief Title: Therapeutic Vaccination and Immune Modulation - New Treatment Strategies for the MDR Tuberculosis Pandemic
Acronym: TBCOX2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anne Margarita Dyrhol Riise (Other)
Collaborators: University of Oslo (Other); Statens Serum Institut (Other); Haukeland University Hospital (Other)
Responsible Party: Sponsor-Investigator, Anne Margarita Dyrhol Riise, Professor, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/692; 2014-004986-26 (EudraCT Number)
Record Dates: First submitted 2015-07-10; First posted 2015-07-21 (Estimated); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Tuberculosis
Keywords: Host-modulating therapy; Vaccine; Cyclooxygenase inhibitors
MeSH Terms: conditions — Tuberculosis | interventions — Etoricoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm#1 (Experimental): arm#1 (n=10) receiving etoricoxib from inclusion day 0 and in 140 days.
  Step-wise inclusion starting with arm#1,arm#2 and arm#3 (first group) randomized (2:2:1) and if safety data are satisfactory proceeding with arm #4 and the rest of arm#3 randomized (2:2:1).
  Interventions: Drug: etoricoxib
- Arm#2 (Experimental): arm#2 (n=10) receiving H56:IC31 vaccine at day 84 and 140 and no etoricoxib.
  Interventions: Biological: H56:IC31
- Arm#3 (No Intervention): arm#3 (n=10), the first group (n=5) serving as control to arm#1 and arm#2, the next group (n=5) serving as control to arm#4.
- Arm#4 (Experimental): arm#4 (n=10) receiving etoricoxib from inclusion day 0 and in 140 days and H56:IC31 vaccine at day 84 and 140.
  Interventions: Drug: etoricoxib; Biological: H56:IC31

INTERVENTIONS:
Drug: etoricoxib — cyclooxygenase-2 inhibitor. Anti-inflammatory
  Other Names: Arcoxia®
  Arms: Arm#1; Arm#4
Biological: H56:IC31 — Therapeutic and prophylactic TB vaccine
  Arms: Arm#2; Arm#4

SUMMARY:
Tuberculosis (TB) is a global challenge and for the increasing epidemic of multi-drug resistant (MDR)-TB there is restricted treatment options. This calls for research of new immune-modulating treatment strategies that can strengthen the patients immune system to better fight the TB bacteria. The pro-inflammatory, but still immunosuppressive mediator prostaglandin E2 (PGE2) is produced by cyclooxygenase-2 (COX-2) in inflamed infected tissue. Studies from both human and animal models show that COX-2 inhibitors (COX-2i) can improve the immune system and strengthen vaccines responses.

Hypothesis

1. A hyperactive COX-2/PGE2 signal system in active TB causes down-regulated immune responses that favour TB survival, but this can be abrogated by COX-2i.
2. TB-specific immunisation with targeted antigens presented as a therapeutic TB vaccine and enhanced by COX-2i will improve immune-mediated host clearance of TB.
3. Combinations of COX-2i and a therapeutic TB vaccine to conventional anti-TB chemotherapy offer new treatment modalities for TB, including MDR/XDR-TB.

Approach to test the hypothesis

1. Study design: 4-arm, open and randomized clinical intervention trial of patients starting treatment for active TB in specialized Norwegian TB centres and where two arms will receive the COX-2i etoricoxib with and without a TB vaccine, one arm vaccine only and the last arm serve as control receiving only standard anti-TB therapy. For safety precautions, only patients bearing sensitive TB strains are included and study arms will be sequentially introduced.
2. In a mouse model examine in more detail the effects of reversion of chronic inflammation with COX-2i locally in tissue and the interplay with TB vaccine responses, immune regulation, correlates of protection and survival in a well-characterized model for TB-exposed mice.

DETAILED DESCRIPTION:
The hypothesis is that treating TB patients with a therapeutic TB vaccine and COX-2 inhibiting drugs in addition to standard antibiotic TB therapy will improve the patients immune system and boost TB vaccine responses.

The project will provide safety and immunogenicity data from a Norwegian phase 1 clinical trial of the therapeutic TB vaccine candidate H56:IC31 and the COX-2i etoricoxib given to TB patients together with standard TB antibiotics.

The investigators will also perform exploratory in-depth studies of immune regulatory mechanisms and try to identify biomarkers for efficacy of treatment both in humans and in a parallel mouse model. These results may further optimize the therapeutic strategy and prepare for larger clinical trials and finally contribute to new treatment options for MDR-TB.

Objectives:

* Study the safety and tolerability of etoricoxib given for 20 weeks (day 0-140) alone and in combination with the therapeutic TB vaccine H56:IC31 given as two immunizations at day 84 and day 140 in patients with active TB disease treated with conventional 26-week anti-TB chemotherapy.
* Study the immune effects of etoricoxib given for 20 weeks (day 0-140) on immune regulation and TB vaccine (H56:IC31) immunogenicity in patients with active TB disease treated with conventional 26-week anti-TB chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 70 years at the time of randomization.
2. Microbiologically confirmed pulmonary TB (culture and/or PCR + susceptibility testing) and/or microbiologically confirmed extra-pulmonary TB (culture and/or PCR + susceptibility testing).
3. Drug sensitive Mtb strains (except single resistance where fully adequate anti-TB chemotherapy regimen could be provided).
4. Is willing and likely to comply with the trial procedures and is prepared to grant authorized persons access to their medical record.
5. Has completed the written informed consent process prior to the start of screening evaluations.
6. Females: Ability to avoid pregnancy during the trial.

Subjects may receive H56:IC31 vaccination (arm#2 and #4) if they meet the following criteria:

1. Sputum obtained prior to 1th immunization (day 84) must be Mtb negative evaluated by at least two consecutive AFS or GeneXpert/PCR at least 7 days apart.
2. Documented reduction in the extent of TB disease at the infectious site(s) within day 84 evaluated by physical and/or radiological examination.
3. Clinical improvement with normal vital signs (blood pressure, temperature and pulse), improvement of any TB related symptoms to Grade 1-3, stable or increased body-weight and reduced inflammatory blood parameters (CRP, ESR and WBC counts) compared to baseline.

Exclusion Criteria:

Main exclusion criteria:

(i) Study-specific: Disseminated TB. Evidence of a new acute illness that may compromise the safety of the subject in the trial on study day 0. History of autoimmune disease or immunosuppression. History or laboratory evidence of any possible immunodeficiency state. Anemia (<9 g/100 ml). HIV sero-positivity. Chronic hepatitis B (HBs antigen positive) with increased liver transaminases (ASAT, ALAT) or chronic hepatitis C (HCV RNA positive). Concomitant or sporadic use of NSAID or corticosteroids (>2 times per week). Other immune modulating therapies including DMARDS. Total cholesterol > 7 mmol/L. Hypertension >140/90 mm Hg (treated or untreated) or treated with >1 antihypertensive drug at any blood pressure. Cardiovascular events or stroke in parents, siblings or off-springs occurring < 55 years of age. Serum creatinine above reference levels (females > 90 µmol/L; males > 105 µmol/L). Known diabetes mellitus type I or diabetes mellitus type II with HbA1c >7%. Pregnancy (S-hCG >5 IU/l for females at childbearing age). Breastfeeding.

2. Exclusion criteria for etoricoxib according to SPC: Known hypersensitivity for etoricoxib or etoricoxib tablet substances. Known hypersensitivity for sulphonamides. Active peptic ulcer or gastrointestinal haemorrhage. History of asthma, acute rhinitis, nasal polyps, angioneurotic oedema, urticaria or other allergic reactions after taking acetyl salicylic acid or NSAID including COX-2 inhibitors. Moderate/severe deranged liver function (Child-Pugh >7). Serum-creatinine clearance < 30 ml/min. Inflammatory bowel disease. Heart failure (NYHA II-IV). Established ischaemic heart disease, peripheral arteriosclerosis and/or cerebrovascular disease, including previous myocardial infarction, angina pectoris, unstable angina, PCI or coronary bypass, previous transitory ischemic attack or apoplexia/stroke.

3. Exclusion criteria for H56:IC31: Known hypersensitivity for vaccines or vaccine adjuvants.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Safety of etoricoxib (arm#1) assessed by the number of participants with adverse events | From day 0 until day 238 (14 weeks after the last dose of etoricoxib)
  Number and % of study patients with AE or SAE
Safety of H56:IC31 vaccine (arm#2) assessed by the number of participants with adverse events | From day 0 until day 238. For vaccine related adverse events; immunisation (day 84 and day 140) and 14 days post-immunisation (day 98 and day 154).
  Number and % of study patients with AE or SAE
Safety of combined etoricoxib and H56:IC31 vaccine (arm#4) assessed by the number of participants with adverse events | From day 0 until day 238 (14 weeks after the last dose of etoricoxib). For vaccine related adverse events; from immunisation (day 84 and day 140) and 14 days post-immunisation (day 98 and day 154).
  Number and % of study patients with AE or SAE
Immunogenicity of etoricoxib (arm#1) | Day 0 (baseline) to day 84
  Total CD4+ T cell cytokine (IFN-γ, IL-2, TNF-α) responses to sum TB peptides.
Immunogenicity of H56:IC31 vaccine (arm#2) | From before first immunisation (day 84) to 14 days after second immunisation (day 154).
  Total CD4+ T cell cytokine (IFN-γ, IL-2, TNF-α) responses to sum TB peptides.
Immunogenicity of combined etoricoxib and H56:IC31 vaccine (arm#4) | From before first immunisation (day 84) to 14 days after second immunisation (day 154).
  Total CD4+ T cell cytokine (IFN-γ, IL-2, TNF-α) responses to sum TB peptides.

SECONDARY OUTCOMES:
Exploratory immune studies | From day 0 (baseline) until day 238 (study end); 14, 28, 56, 84, 98, 140, 154, 182, 210, 238 days from baseline (selected timepoints for various analysis).
  Study in depth the effect of etoricoxib on immune activation, regulation and TB vaccine immunogenicity measured by the percentage of innate cells (monocytes/MDSC) and CD4+ and CD8+ T cells expressing various activation, supression and regulation markers in response to stimulation with TB antigenic peptide pools (Ag85B, ESAT-6, Rv2660c). Serologi to H56 and gene signature analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Margarita Dyrhol-Riise, PhD, Principal Investigator — Oslo University Hospital
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: Yes
The study is published. https://doi.org/10.1038/s41467-021-27029-6
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data available as supplementary information in the published manuscript.
Access Criteria: The full source datasets generated during and/or analyzed during the current study are available in the repository of the open science framework (https://osf.io/khvf4)
URL: https://doi.org/10.1038/s41467-021-27029-6

REFERENCES:
- [Derived] Nore KG, Louet C, Bugge M, Gidon A, Jorgensen MJ, Jenum S, Dyrhol-Riise AM, Tonby K, Flo TH. The Cyclooxygenase 2 Inhibitor Etoricoxib as Adjunctive Therapy in Tuberculosis Impairs Macrophage Control of Mycobacterial Growth. J Infect Dis. 2024 Mar 14;229(3):888-897. doi: 10.1093/infdis/jiad390. PMID 37721470
- [Derived] Jenum S, Tonby K, Rueegg CS, Ruhwald M, Kristiansen MP, Bang P, Olsen IC, Sellaeg K, Rostad K, Mustafa T, Tasken K, Kvale D, Mortensen R, Dyrhol-Riise AM. A Phase I/II randomized trial of H56:IC31 vaccination and adjunctive cyclooxygenase-2-inhibitor treatment in tuberculosis patients. Nat Commun. 2021 Nov 22;12(1):6774. doi: 10.1038/s41467-021-27029-6. PMID 34811370
- [Derived] Tonby K, Mortensen R, Ruhwald M, Dyrhol-Riise AM, Jenum S. KLRG1-Expressing CD4 T Cells Are Reduced in Tuberculosis Patients Compared to Healthy Mycobacterium tuberculosis-Infected Subjects, but Increase With Treatment. J Infect Dis. 2019 Jun 5;220(1):174-176. doi: 10.1093/infdis/jiz056. No abstract available. PMID 30888024

DOCUMENTS (2):
  • Study Protocol (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT02503839/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/39/NCT02503839/SAP_001.pdf